CLINICAL TRIAL: NCT00938418
Title: Phase II Study on Dose Escalated, Accelerated Hypofractionated Intensity Modulated Radiotherapy for Stage III Non-Small Cell Lung Cancer With Concurrent Chemotherapy
Brief Title: Hypofractionated Intensity Modulated Chemoradiotherapy to Treat Locally Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Dr Ivan Tham, National University Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B/09/108
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Stage III Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Radiation: Dose escalated, accelerated, hypofractionated radiotherapy — Intensity modulated radiotherapy with concurrent chemotherapy

SUMMARY:
Locally advanced non-small cell lung cancer can be treated successfully with chemotherapy and radiation. However, the cure rate is low.

This study is carried out to find out whether giving radiotherapy at a higher dose over fewer treatment sessions with intensity modulated radiotherapy (IMRT) can improve the treatment outcome.

This study aims to recruit 43 patients from National University Hospital and Tan Tock Seng Hospital over a period of about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of Stage IIIA or IIIB non-small cell lung cancer; excluding patients with N3 disease based on supraclavicular or contralateral hilar adenopathy, or significant pleural / pericardial effusion.

Exclusion Criteria:

* Patients for whom treatment is planned with a maximum dose of ≥ 66 Gy to the ipsilateral brachial plexus
* Greater than minimal, exudative, or cytologically positive pleural effusions
* ≥ 10% weight loss within the past month
* Prior invasive malignancy (with exceptions)
* Prior radiotherapy to the region of the study cancer
* Significant co-morbidities
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Known allergic reactions to components of planned chemotherapy regimen

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Response rate, locoregional control, disease free survival, toxicity | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore